CLINICAL TRIAL: NCT07015411
Title: Effectiveness of an Orally Administered and Combined Neuro-Complex & Multi Supplements in the Prevention of Migraine in Adult
Brief Title: Neuro-Complex & Multi Supplements for Migraine Prevention
Acronym: NeuroCare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benfida, a department of Handi-Move (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2025-05-19; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Migraine Headache; Migraine; Migraine in Adults
Keywords: Migraine; Neuro-Complex; Multi; Supplement; headache; nutrients
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplementation Arm - Neuro-Complex and Multi Combination (Experimental)
  Interventions: Dietary Supplement: Neuro-Complex and Multi

INTERVENTIONS:
Dietary Supplement: Neuro-Complex and Multi — Participants will orally consume 2 caps of each product (taken at the same time) daily, one in the morning and one at the lunchtime preferably during meal, for 8 weeks after a running period of 8 weeks without supplementation. Intake will be initiated from the day of follow-up visit (V1) after all study procedures being performed until the day of the end-of-study visit (V2).
  Participants will take 1 cap of each product simultaneously twice a day directly in their mouth.

SUMMARY:
The goal of this prospective, monocentric, open-label, non-randomized and single arm study is to evaluate a reduction of migraine days per months (MDM) by 25% by using the combined supplementation with Neuro-Complex & Multi after 8 weeks of product intake on participants with diagnosis of migraine meeting the criteria of the International Classification of Headache Disorders (ICHD-3) (with or without aura).

The main endpoint of this clinical trial is :

The mean changes in migraine days per month (MDM) after 8 weeks of supplementation.

Participants will:

Orally consume two caps of each product (taken at the same time) daily, one in the morning and one at the lunchtime preferably during meal, for 8 weeks after a running period of 8 weeks without supplementation. Intake will be initiated from the day of follow-up visit (V1) after all study procedures being performed until the day of the end-of-study visit (V2).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years;
* Diagnosis of migraine meeting the criteria of the International Classification of Headache Disorders (ICHD-3) (with or without aura)

  * At least 5 attacks fulfilling the criteria below
  * Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)
  * Headache has at least two of the following characteristics

    * unilateral location
    * pulsating quality
    * moderate or severe pain intensity
    * aggravation by or causing avoidance of routine physical activity (eg, walking or climbing stairs)
  * During headache at least one of the following:

    * nausea and/or vomiting
    * photophobia and phonophobia
  * Not attributed to another disorder
* Migraine frequency of at least 6 headache days per month during the last 3 months;
* Stable body mass index (BMI) between 18.5-35.0;
* Stable medication use with no significant changes in prophylactic or acute migraine treatments in the past 3 months, and willingness to maintain or reduce (if not needed) this throughout the study period;
* Willingness and ability to complete an ediary (mobile app or web based) and to follow the instruction of the study;
* Having signed an informed consent.

Exclusion Criteria:

* Other primary head pain disorders such as but not restricted to tension-type headache, cluster headache, fibromyalgia;
* Secondary head pain due to trauma, injury, infections;
* Medication overuse for headache defined as acute headache medication >10-15 days per month depending on the half-life of the medication (left to PI discretion);
* Severe medical conditions affecting absorption and metabolism of the product, including but not restricted to chronic use of laxatives;
* Bariatric surgery;
* Severe psychiatric conditions that could interfere with diary compliance or assessment of the product (e.g., severe depression or cognitive impairments) left to investigator discretion;
* Use of other dietary supplements that could potentially affect migraines, unless willing to discontinue them before the study begins (wash out period of 3 months);
* Women who are pregnant, breastfeeding, or planning to become pregnant during the study period;
* Women of childbearing potential without medically effective form of contraception unless they can confirm they've had bilateral tubal ligation or that their male partner has had a vasectomy;
* Specific allergies or intolerance to components of the product;
* Recent migraine interventions: Such as Botox injections (except if considered as a stable treatment, i.e. not the first injection), nerve blocks, or other invasive treatments in the last 6 months;
* Concurrent participation in another clinical study or having participated in the last 3 months:
* Swallowing disorders;
* Chronic drug and alcohol abuse;
* Anticoagulants (coumarin compound);
* Hepatic or biliar truct disorders;
* Active malignancy and immunosuppression therapy;
* Hypothyroidism;
* Close collaborators of investigational team, of sponsor or of study coordinator;
* Under guardianship or judiciable protection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
Reduction of migraine days per month (MDM) by 25% by using the combined supplementation with Neuro-Complex & Multi after 8 weeks of product intake | Between Week 8 (V1) and Week 16 (after 8 weeks of supplementation)
  Mean change of migraine days per month (MDM)

SECONDARY OUTCOMES:
Evaluate the effect on migraine intensity/severity after 8 weeks of product intake | Between Week 8 (V1) and Week 16 (after 8 weeks of supplementation)
  Mean change in migraine intensity/severity measured using a numerical rating scale after 8 weeks of product intake
Evaluate the effect on migraine duration after 8 weeks of product intake | Between Week 8 (V1) and Week 16 (after 8 weeks of supplementation)
  Mean change in migraine duration defined as start date and end date of each migraine episode captured by the patient
Evaluate the effect on symptoms associated with migraine after 8 weeks of product intake | Between Week 8 (V1) and Week 16 (after 8 weeks of supplementation)
  Mean change in symptoms measured using a 5-likert scale
Evaluate the effect on quality of life (QoL) after 8 weeks of product intake | Between Week 8 (V1) and Week 16 (after 8 weeks of supplementation)
  Mean change in QoL assessed using self-reported questionnaire (SF-36)
Evaluate the effect on number of responders to the supplementation after 8 weeks of product intake | Between Week 8 (V1) and Week 16 (after 8 weeks of supplementation)
  Proportion of responders defined as patients with ≥50% reduction in MDM
• Evaluate the effect on reduction in the use of acute medication for migraine after 8 weeks of product intake | Between Week 8 (V1) and Week 16 (after 8 weeks of supplementation)
  Mean change in days of use of acute medication against migraine
Evaluate the effect on patient tolerance after 8 weeks of product intake | Between Week 8 (V1) and Week 16 (after 8 weeks of supplementation)
  Mean change in number of Adverse events (AE)
Evaluate the effect on migraine days per month (MDM) after 16 weeks (8 weeks without supplementation followed by 8 weeks of supplementation) | Between Baseline (V0) and Week 16 (after 8 weeks of non-supplementation followed by 8 weeks of supplementation)
  Mean change of migraine days per month (MDM)
Evaluate the effect on migraine intensity/severity after 16 weeks (8 weeks without supplementation followed by 8 weeks of supplementation) | Between Baseline (V0) and Week 16 (after 8 weeks of non-supplementation followed by 8 weeks of supplementation)
  Mean change in migraine intensity measured using a numerical rating scale
Evaluate the effect on migraine duration after 16 weeks (8 weeks without supplementation followed by 8 weeks of supplementation) | Between Baseline (V0) and Week 16 (after 8 weeks of non-supplementation followed by 8 weeks of supplementation)
  Mean change in migraine duration defined as start date and end date of each migraine episode captured by the patient
Evaluate the effect on symptoms associated with migraine after 16 weeks (8 weeks without supplementation followed by 8 weeks of supplementation) | Between Baseline (V0) and Week 16 (after 8 weeks of non-supplementation followed by 8 weeks of supplementation)
  Mean change in symptoms measured using a 5-likert scale
Evaluate the effect on quality of life (QoL) after 16 weeks (8 weeks without supplementation followed by 8 weeks of supplementation) | Between Baseline (V0) and Week 16 (after 8 weeks of non-supplementation followed by 8 weeks of supplementation)
  Mean change in QoL assessed using self-reported questionnaire (SF-36)
Evaluate the effect on number of responders to the supplementation after 16 weeks (8 weeks without supplementation followed by 8 weeks of supplementation) | Between Baseline (V0) and Week 16 (after 8 weeks of non-supplementation followed by 8 weeks of supplementation)
  Proportion of responders defined as patients with ≥50% reduction in MDM
Evaluate the effect on reduction in the use of acute medication for migraine after 16 weeks (8 weeks without supplementation followed by 8 weeks of supplementation) | Between Baseline (V0) and Week 16 (after 8 weeks of non-supplementation followed by 8 weeks of supplementation)
  Mean change in days of use of acute medication against migraine
Evaluate the effect on patient tolerance after 16 weeks (8 weeks without supplementation followed by 8 weeks of supplementation) | Between Baseline (V0) and Week 16 (after 8 weeks of non-supplementation followed by 8 weeks of supplementation)
  Mean change in number of Adverse events (AE)
Compare the effect on migraine days per month (MDM) between the non-supplementation period (baseline to 8 weeks) and the supplementation period (8 to 16 weeks) | Between the non-supplementation period (Baseline to Week 8) and the supplementation period (Week 8 to Week 16)
  Mean change of migraine days per month (MDM)
Compare the effect on migraine intensity/severity between the non-supplementation period (baseline to 8 weeks) and the supplementation period (8 to 16 weeks) | Between the non-supplementation period (Baseline to Week 8) and the supplementation period (Week 8 to Week 16)
  Mean change in migraine intensity measured using a numerical rating scale
Compare the effect on migraine duration between the non-supplementation period (baseline to 8 weeks) and the supplementation period (8 to 16 weeks) | Between the non-supplementation period (Baseline to Week 8) and the supplementation period (Week 8 to Week 16)
  Mean change in migraine duration defined as start date and end date of each migraine episode captured by the patient
Compare the effect on symptoms associated with migraine between the non-supplementation period (baseline to 8 weeks) and the supplementation period (8 to 16 weeks) | Between the non-supplementation period (Baseline to Week 8) and the supplementation period (Week 8 to Week 16)
  Mean change in symptoms measured using a 5-likert scale
Compare the effect on quality of life (QoL) between the non-supplementation period (baseline to 8 weeks) and the supplementation period (8 to 16 weeks) | Between the non-supplementation period (Baseline to Week 8) and the supplementation period (Week 8 to Week 16)
  Mean change in QoL assessed using self reported questionnaire (SF-36)
Compare the effect on number of responders to the supplementation between the non-supplementation period (baseline to 8 weeks) and the supplementation period (8 to 16 weeks) | Between the non-supplementation period (Baseline to Week 8) and the supplementation period (Week 8 to Week 16)
  Proportion of responders defined as patients with ≥50% reduction in MDM
Compare the effect on reduction in the use of acute medication for migraine between the non-supplementation period (baseline to 8 weeks) and the supplementation period (8 to 16 weeks) | Between the non-supplementation period (Baseline to Week 8) and the supplementation period (Week 8 to Week 16)
  Mean change in days of use of acute medication against migraine
Compare the effect on patient tolerance between the non-supplementation period (baseline to 8 weeks) and the supplementation period (8 to 16 weeks) | Between the non-supplementation period (Baseline to Week 8) and the supplementation period (Week 8 to Week 16)
  Mean change in number of Adverse events (AE)

CONTACTS AND LOCATIONS:
Locations (1):
- Meclinas, Mechelen, Belgium